CLINICAL TRIAL: NCT06841588
Title: The Effect of Mulligan's Mobilization with Movement Versus Dry Needling on Pain, Function, and Range of Motion Among Athletes with Hip Adductor Related Groin Pain and Dysfunction
Brief Title: The Effect of Mulligan's Mobilization with Movement Versus Dry Needling on Pain,Function,and Range of Motion Among Athletes with Hip Adductor Related Groin Pain and Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Quds University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 118/REC/2020
Record Dates: First submitted 2025-01-20; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2023-06

CONDITIONS: Hip Adduction Strength; Groin Pain; Groin Injury
Keywords: Athletes; hip adductor; groin pain; athletes with groin pain; athletes with hip dysfunction
MeSH Terms: interventions — Movement; Dry Needling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mulligan's Mobilization with Movement and Dry Needling (Active Comparator): the intervention group 1 was treated using Mulligan Mobilization with Movements and Dry Needling (DN&MWM) for soft tissue trigger points, (N=15).
  Interventions: Other: Mulligan's Mobilization with Movement and Dry Needling
- Dry Needling (Active Comparator): the intervention group 2 was treated using Dry Needling (DN) for soft tissue trigger points, (N=15).
  Interventions: Other: Dry Needling (DN)

INTERVENTIONS:
Other: Mulligan's Mobilization with Movement and Dry Needling — the intervention group 1 was treated using Mulligan Mobilization with Movements and Dry Needling (DN&MWM) for soft tissue trigger points, (N=15).
  The treatment duration was 6 sessions, 3 sessions per week ( day after day).
  Arms: Mulligan's Mobilization with Movement and Dry Needling
Other: Dry Needling (DN) — The intervention group 2 was treated using Dry Needling (DN) for soft tissue trigger points, (N=15). The treatment duration was 6 sessions, 3 sessions per week ( day after day).
  Arms: Dry Needling

SUMMARY:
This study aims to highlight and investigate the effectiveness of two common management practices in physiotherapy, dry needling intervention as a soft tissue technique and Mulligan mobilization with movements MWM as a joint technique, on pain, function, and range of motion among athletes with hip adductor-related groin pain and dysfunction.

DETAILED DESCRIPTION:
Background:

Injuries are considered a common challenge in the sports field, 31% of the injuries are muscular, especially in the lower extremities. Injuries in the groin area are a major and serious problem because they are common, lead to prolonged symptoms, and had a high recurrence rate.

Study objective:

This study aims to highlight and investigate the effectiveness of two common management practices in physiotherapy, dry needling DN intervention as a soft tissue technique and Mulligan mobilization with movements MWM as a joint technique.

Methods:

A convenience sampling of thirty football players who were diagnosed with hip adductor-related groin pain and dysfunction were recruited from different cities in the west bank who participated in this randomized clinical trial, the participants were randomly divided into two groups, the dry needling group (15), and dry needling combined with Mulligan mobilization MWM (15).

Numiric Pain Rating Scale (NPRS), Five-Second Copenhagen Squeeze test, Hip Abduction Range of Motion, Adductor Squeeze Test, Flexion Abduction External Rotation Test (FABER), Y Balance Test, and The Copenhagen Hip and Groin Outcome Score (HAGOS) were used as outcome measures (NPRS and 5-second squeeze test performed each session for the two groups).

ELIGIBILITY:
Inclusion Criteria:

1. Athletes suffered from unilateral adductor-related groin pain, grades 1 and 2.
2. Acute, subacute, or chronic athletes with hip adductor-related groin pain and dysfunction.
3. Groin pain during or after activities.
4. Pain at palpation of the adductors and their origin.
5. Pain on resistance against adduction.
6. Aged 15- 35 years old.

Exclusion criteria:

Patients with other causes of groin pain such as:

1. Lymphadenitis.
2. Prostatitis, Urinary infections, Malignancy.
3. Spinal pathology.
4. Hip joint osteoarthritis.
5. Inguinal-related or Iliopsoas-related groin pain.
6. Femoral or Inguinal hernia.
7. Referral pain and adductor strain grade 3.
8. Current use of medication.

Ages: 15 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Athletes males
Enrollment: 30 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Sheet of Demographic Data | pre and 1 day post treatment
  Demographic, personal data, and injury history were obtained at baseline from the patient interview and recorded on a data collection sheet
Numeric Pain Rating Scale NPRS | pre and 1 day post treatment
  The Numeric Pain Rating Scale (NPRS) is valid and reliable, a self-assessing questionnaire , used to assess the severity of pain. 0- 10 scale where 0 represents "no pain" and 10 representing "unbearable pain." Each participant was asked to indicate the pain level before and after treatment.
Y-Balance Test YBT | pre and 1 day post treatment
  The Y balance test was developed from the star excursion balance test (SEBT) and assesses performance during single-leg balance with reaching in the 3 directions: anterior, posteromedial, and posterolateral. the patient stands on one leg while reaching out in 3 different directions with the other lower extremity.
FABER Test | pre and 1 day post treatment
  To assess the adductor muscle tightness and shortening due to injury. FABER test is used as a provocation special test but has also been used as a measurement of combined hip range of motion, also useful tools for the hip examination, particularly for anterior hip or groin pain. The patient lies supine on the examination table. The hip and knee of the tested leg are flexed, abducted, and externally rotated, as the foot of the tested leg is placed on the contralateral thigh just proximal to the knee. While stabilizing the pelvis on the contralateral side, gentle pressure is applied downwards on the knee of the tested leg, also measuring the distance from the lateral condyle of the knee to the surface of the examination table for both affected and none affected knees.
Five Seconds Copenhagen Squeeze Test | pre and 1 day post treatment
  The therapist placed his arms between the athlete's knees and asked the athlete to squeeze the legs as hard as possible for five seconds, then, scored any pain in the groin area on a scale of 0 to 10 NPRS Scale

CONTACTS AND LOCATIONS:
Overall Officials: Daragmah, Master degree, Principal Investigator — Al-Quds University
Locations (1):
- Ayman Daragmah, Ramallah, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No